CLINICAL TRIAL: NCT06278376
Title: Evaluation of Diagnoses and Clinical Outcomes in Children Undergoing MRI Scans: a Retrospective, Longitudinal Study
Brief Title: Evaluation of Diagnoses and Clinical Outcomes in Children Undergoing MRI Scans
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Professor Anesthesiology, MD, PhD, Jessa Hospital
Other Study IDs: f/2023/045
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Magnetic Resonance Imaging
Keywords: Magnetic Resonance Imaging; Childeren

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to evaluate the indications and therapeutical consequences of MRI scans of (young) children undergoing risky remote anaesthesia. The investigators want to aim for a clear indication in children undergoing MRI in the future before undergoing possible unnecessary procedures and MRI scans.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is a non-invasive imaging technique that allows physicians to visualize our anatomy, generating high-quality pictures of our body's internal structure at many different angles. The principle behind MRI, known as nuclear magnetic resonance (NMR), revolves around hydrogen atoms (or protons) that can be found everywhere in our entire body, such as in bones, blood, organs, skin, muscles and more. Protons have their own magnetic moment and angular momentum, allowing them to spin in a certain direction. By subjecting these spinning protons to a strong magnetic field they will be oriented along the axis of the magnetic field, either with or against the direction of the magnetic field. MRI machines generate this field using a large magnet surrounding the patient. Electric gradient coils allow the strength of the field to be adjustable, usually around 0,5 or 1,5 tesla.

MRI has many advantages compared to other imaging techniques, i.e. CT (computed tomography), including the lack of radiation, the ability to show abnormalities of soft tissues, the ability to visualize blood flow, and contrasting agents that are less likely to cause adverse effects like allergic reactions. There are also some disadvantages or limitations, however: implants or metallic objects inside the body can make images unclear at best or harm the patient at worst; similarly, movements made by the patient can make images unclear as well. Lastly, MRI is a more expensive and slower technique compared to other imaging techniques.

Children undergoing an MRI are often sedated before being placed inside the machine. After the scan is over, the children will be brought to a recovery area, where they can slowly recover from the sedation until they are fully awake again. Some common side effects resulting from the sedation may be vomiting, drowsiness and/or dizziness.

The aim of this study is to evaluate the indications and therapeutical consequences of MRI scans of (young) children undergoing risky remote anaesthesia. The investigators want to aim for a clear indication in children undergoing MRI in the future before undergoing possible unnecessary procedures and MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing an MRI scan in Jessa hospital (Hasselt, Belgium) between November 2016 and February 2023.
* Age between 6 months and 16 years

Exclusion Criteria:

* /

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population for this study will be children between 6 months and 16 years old who have undergone an MRI scan in Jessa hospital (Hasselt, Belgium) between November 2016 and February 2023.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence | Between 2016 and 2023
  Incidence of diagnostic MRI in childeren

SECONDARY OUTCOMES:
Therapeutical implications: diagnosis | Between 2016 and 2023
  Evaluating the presence of a diagnosis after this MRI investigation
Therapeutical implications: treatment | Between 2016 and 2023
  Evaluating if the MRI investigation resulted in treatment (drug treatment, surgery or physiotherapy)
Clinical indications | Between 2016 and 2023
  Evaluating the clinical indications for the MRI investigation
Evaluation of body part | Between 2016 and 2023
  Evaluating which specific body parts are undergoing imaging
Evaluation of symptoms | Between 2016 and 2023
  Evaluation of the pre-existing symptoms (vomiting, headache, developmental delay, sleep issures, swellings, seizures, balance problems, conduct disorders, febrile convulsions) that potentially lead to an MRI scan
Clinical outcome: adverse event | Between 2016 and 2023
  Evaluation of the clinical outcome: adverse events
Clinical outcome: surgery | Between 2016 and 2023
  Evaluation of the clinical outcome: surgery after MRI
Clinical outcome: admission to hospital | Between 2016 and 2023
  Evaluation of the clinical outcome: admission to hospital
Clinical outcome: mortality | Between 2016 and 2023
  Evaluation of the clinical outcome: mortality after MRI
Evaluation of age | Between 2016 and 2023
  Evaluation of age in children: <2 years, 2-6 years and >6 years
Influence of COVID-19 pandemic | Between 2016 and 2023
  Influence of COVID-19 pandemic (2020-2021 versus 2016-2017-2018-2019-2022-2023) on incidence, therapeutical implications and outcomes of MRI scans in children

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No